CLINICAL TRIAL: NCT06134388
Title: Clinical Study Evaluating the Efficacy and Safety of Sulfasalazine in Patients With Metastatic Colorectal Cancer
Brief Title: Sulfasalazine in Patients With Metastatic Colorectal Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Reham Ameen El-Ghoneimy, Assistant Lecturer of Clinical Pharmacy, Faculty of Pharmacy, Tanta University, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sulfasalazine 2023
Record Dates: First submitted 2023-11-05; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Sulfasalazine; mCRC
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Sulfasalazine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): This group will include 25 patients who will be scheduled to receive 6 cycles of 5-Fluorouracil and Oxaliplatin- based regimens every 2 weeks for 3 months.
- Sulfasalazine Group (Active Comparator): This group will include 25 patients who will be scheduled to receive 6 cycles of 5-Fluorouracil and Oxaliplatin- based regimens every 2 weeks plus sulfasalazine (1 gram orally twice daily) for 3 months.
  Interventions: Drug: Sulfasalazine

INTERVENTIONS:
Drug: Sulfasalazine — Sulfasalazine is an anti-inflammatory drug that is indicated for treatment of ulcerative colitis and rheumatoid arthritis.
  Arms: Sulfasalazine Group

SUMMARY:
The aim of this study is to evaluate the potential efficacy and safety of sulfasalazine in patients with metastatic colorectal cancer.

DETAILED DESCRIPTION:
Sulfasalazine is an anti-inflammatory drug that is indicated for treatment of ulcerative colitis and rheumatoid arthritis. Sulfasalazine decreased the risk of ulcerative colitis-related colorectal cancer through its anti-inflammatory effect and induction of oxidative stress in cancer cells. Furthermore, intact sulfasalazine, but not its metabolites, inhibited the growth and metastasis various cancers.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of stage IV (metastatic) colorectal cancer. Staging will be performed according to the American Joint Committee on Cancer (AJCC) 8th edition and will be documented by all investigating parameters of metastatic colorectal cancer
2. Male or female patients with age range from 18-65 years old
3. Women of childbearing age will be required to be on acceptable forms of contraception
4. Performance status < 2 according to the Eastern Cooperative Oncology Group (ECOG) score
5. No contraindication to chemotherapy (absence of myelosuppression)
6. Adequate liver function (alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < grade 2) according to the National Cancer Institute-Common Terminology Criteria for Adverse Events, version 5.0 (NCI-CTCAE v 5.0)
7. Adequate renal function (estimated creatinine clearance (eCrCl), serum creatinine (SCr) < grade 2) according to NCI-CTCAE, v 5.0
8. Adequate hematological parameters (hemoglobin, erythrocytes, platelets, leukocytes and absolute neutrophil count (ANC) < grade 2 according to NCI-CTCAE, v 5.0

Exclusion Criteria:

1. Pregnant or lactating women
2. Patients with concurrent active cancer originating from a primary site other than the colon or rectum
3. Patients who have known allergy to sulfasalazine or its metabolites
4. Patients with nephrolithiasis, severe vomiting or severe diarrhea
5. Patients who are receiving highly plasma protein-bound drugs or drugs with extensive hepatic metabolism such as; coumarin anti-coagulants
6. Patients with intestinal or urinary obstruction
7. Patients with known glucose-6-phosphate dehydrogenase deficiency or porphyria
8. Ongoing treatment with sulfasalazine or mesalamine for ulcerative colitis or rheumatoid arthritis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Evaluating the change in the serum level of Ferritin | 3 months
  Blood samples will be collected at baseline and 3 months after treatment.
Evaluating the change in the serum level of Superoxide dismutase (SOD) | 3 months
  Blood samples will be collected at baseline and 3 months after treatment.
Evaluating the change in the serum level of Nuclear factor-kappa B (NF-kB) | 3 months
  Blood samples will be collected at baseline and 3 months after treatment.
Evaluating the change in the serum level of Bcl-2 associated X protein (Bax) | 3 months
  Blood samples will be collected at baseline and 3 months after treatment.
Investigating the possible efficacy of sulfasalazine through evaluation of its impact on overall response rate (ORR). | 3 months
  Abdominal, pelvic and chest CT scanning will be performed at baseline and after 3 months. ORR will be evaluated and categorized according to the RECIST 1.1 criteria. ORR includes patients with both complete response and partial response. ORR will be determined as number and percentage.
Investigating the possible efficacy of sulfasalazine through evaluation of its impact on disease control rate (DCR). | 3 months
  Abdominal, pelvic and chest CT scanning will be performed at baseline and after 3 months. DCR will be evaluated and categorized according to the RECIST 1.1 criteria. DCR includes patients with complete response, partial response and stable disease. DCR will be determined as number and percentage.

SECONDARY OUTCOMES:
Evaluating the progression free survival (PFS) | 12 months
  PFS is defined as the time from randomization to investigator- assessed tumor progression. PFS will be determined as mean and median in months.
Evaluating the one-year overall survival (1-year OS) | 12 months
  OS is defined as the time from randomization to death from any cause is OS. One-year OS will be determined as mean and median in months.
Evaluating the safety and tolerability of sulfasalazine through investigating Hematological parameters (hemoglobin (mg/dL), erythrocytes (cells/μL), leukocytes (cells/μL), platelets (cells/μL) and absolute neutrophil count (cells/μL)). | 3 months
  These parameters will be followed up at baseline and 3 months after treatment. The reported adverse effects will be graded according to the National Cancer Institute- Common Terminology Criteria for Adverse Effects ( NCI-CTCAE) version 5.
Evaluating the safety and tolerability of sulfasalazine through investigating Liver function test. | 3 months
  These parameters will be followed up at baseline and 3 months after treatment. The reported adverse effects will be graded according to the National Cancer Institute- Common Terminology Criteria for Adverse Effects ( NCI-CTCAE) version 5.
Evaluating the safety and tolerability of sulfasalazine through investigating Renal function test (serum creatinine (mg/dL), blood urea nitrogen (mg/dL) and creatinine clearance (mL/min)). | 3 months
  These parameters will be followed up at baseline and 3 months after treatment. The reported adverse effects will be graded according to the National Cancer Institute- Common Terminology Criteria for Adverse Effects ( NCI-CTCAE) version 5.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University Hospital, Tanta, El-Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ma MZ, Chen G, Wang P, Lu WH, Zhu CF, Song M, Yang J, Wen S, Xu RH, Hu Y, Huang P. Xc- inhibitor sulfasalazine sensitizes colorectal cancer to cisplatin by a GSH-dependent mechanism. Cancer Lett. 2015 Nov 1;368(1):88-96. doi: 10.1016/j.canlet.2015.07.031. Epub 2015 Aug 5. PMID 26254540
- [Background] Yin L, Liu P, Jin Y, Ning Z, Yang Y, Gao H. Ferroptosis-related small-molecule compounds in cancer therapy: Strategies and applications. Eur J Med Chem. 2022 Dec 15;244:114861. doi: 10.1016/j.ejmech.2022.114861. Epub 2022 Oct 22. PMID 36332549
- [Background] Narang VS, Pauletti GM, Gout PW, Buckley DJ, Buckley AR. Sulfasalazine-induced reduction of glutathione levels in breast cancer cells: enhancement of growth-inhibitory activity of Doxorubicin. Chemotherapy. 2007;53(3):210-7. doi: 10.1159/000100812. Epub 2007 Mar 15. PMID 17356269